CLINICAL TRIAL: NCT01835587
Title: A Phase 1/2 Dose and Schedule Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Oral Azacitidine (CC-486) in Subjects With Acute Myelogenous Leukemia and Myelodysplastic Syndromes After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Safety Study of Oral Azacitidine (CC-486) as Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) in Participants With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes (MDS).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-AML-002
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: Acute myeloid leukemia,; myelodysplastic syndromes,; CC-486, oral Azacitidine,; transplantation,; allogeneic,; HSCT.
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-486 (Experimental): Dose of 150 mg, 200 mg, or 300 mg once daily (QD) for the first 7, 10, or 14 days of each 28-day cycle, starting 42-84 days after transplantation.
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: CC-486 — Cohorts of 3 to 6 subjects will be treated at escalating or de-escalating sequential dose levels until a preliminary Maximum Tolerated Dose (MTD) is identified.
  Other Names: Oral Azacitdine

SUMMARY:
The purpose of the study is to determine the maximal tolerated dose and schedule of CC-486, known as oral azacitidine, in patients with AML or MDS after allogeneic hematopoetic stem cell transplant (HSCT). HSCT is more frequently used in AML or MDS as a potential curative therapy. However, disease recurrence/relapse and graft-versus-host disease (GVHD) remain the principal causes of fatal complications after transplantation. Oral azacitidine has significant activity in MDS and AML. Oral azacitidine has also demonstrated immunomodulatory activity in AML patients after allogeneic HSCT. An oral formulation of oral azacitidine provides a convenient route of administration and an opportunity to deliver the drug over a prolonged schedule.

DETAILED DESCRIPTION:
This is an open-label, multicenter study of oral azacitidine in MDS or AML patients who have undergone allogeneic HSCT. The study consists of three phases: Screening, Treatment and Follow-up. During the Screening phase, the study doctor will do tests to see if the patient is suitable for this study. The patients meeting protocol-specified entry criteria will enter the treatment phase and be assigned to receive one of the oral azacitidine cohorts. The dosing group of 200 mg QD on Days 1 to 7 will be evaluated first (ie, Cohort 1). In the event that unacceptable toxicity occurs in Cohort 1, then oral azacitidine may be evaluated at lower dose levels (eg, 150 mg). If the dosing regimen is confirmed to be safe in Cohort 1, other cohorts will be evaluated sequentially. During the treatment phase, patients will be monitored closely for safety and tolerability. Dosing interruption or delay, dose or schedule reduction, intra-subject dose/schedule escalation or re-escalation may occur on the basis of protocol-specified dosing adjustment guidelines. Safety will be monitored throughout the study at predetermined intervals and as clinically indicated by vital signs, physical examination, performance status, laboratory tests and evaluation of adverse events. The patient can continue to receive the study treatment for up to 12 months provided that they benefit from the study treatment and all protocol-specified criteria are met. However, the patient may receive the study treatment for less than 12 months due to adverse event, disease recurrence or progression. When the study treatment is discontinued, all patients who have received at least one dose of oral azacitidine will be asked to see the study doctor for the treatment discontinuation visit. Thereafter, all patients discontinued from the study treatment will enter the Follow-up phase for safety and survival follow up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Myelodysplastic Syndromes or Acute Myeloid Leukemia undergoing allogeneic hematopoietic stem cell transplantation with either peripheral blood or bone marrow as the source of hematopoietic stem cells

At the time of allogeneic HSCT:

* No prior allogeneic HSCT; and
* No more than 1 antigen mismatch at Human Leukocyte Antigen (HLA)-A, -B, -C, -DRB1 or -DQB1 locus for either related or unrelated donor; and
* Bone marrow blast < 20% if MDS or ≤ 10% if AML; and
* Peripheral blood blast ≤ 5%

Be able to start study drug between 42 to 84 days following allogeneic HSCT

Post transplant bone marrow blast count ≤ 5% confirmed within 21 days prior to starting study therapy

Adequate engraftment within 14 days prior to starting study therapy:

* Absolute Neutrophil count (ANC) ≥ 1.0 x 10^9/L without daily use of myeloid growth factor; and
* Platelet count 75 x 10^9/L without platelet transfusion within one week.

Adequate organ function:

* Serum aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
* Serum bilirubin < 2 x ULN
* Serum creatinine < 2 x ULN

Adequate coagulation (Prothrombin time [PT] ≤ 15 seconds, Partial thromboplastin time (PTT) ≤ 40 seconds, and/or International normalized ratio [INR] ≤ 1.5)

Have a negative serum pregnancy test (sensitivity of at least 25 mIU/mL at screening).

Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Must agree to follow protocol-specified pregnancy precautions

Exclusion Criteria:

* Use of any of the following after transplantation and prior to starting oral azacitidine:

  * Chemotherapeutic agents for chemotherapy
  * Investigational agents/therapies
  * Azacitidine, decitabine or other demethylating agents
  * Lenalidomide, thalidomide and pomalidomide

Active Graft-versus-host disease (GVHD) grade II or higher

Any evidence of gastrointestinal (GI) GVHD

Concurrent use of corticosteroids equivalent of prednisone at a dose > 0.5 mg/kg

Known active viral infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV)

Active uncontrolled systemic fungal, bacterial or viral infection

Presence of malignancies, other than MDS or AML, within the previous 12 months

Significant active cardiac disease within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skikne, M.D., FACP; FCP (SA), Study Director — Celgene Corporation
Locations (5):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center., New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MD Anderson Cancer Center The University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Queen Elizabeth Hospital UHB NHS Foundation Trust, Birmingham, United Kingdom

REFERENCES:
- [Derived] de Lima M, Oran B, Champlin RE, Papadopoulos EB, Giralt SA, Scott BL, William BM, Hetzer J, Laille E, Hubbell B, Skikne BS, Craddock C. CC-486 Maintenance after Stem Cell Transplantation in Patients with Acute Myeloid Leukemia or Myelodysplastic Syndromes. Biol Blood Marrow Transplant. 2018 Oct;24(10):2017-2024. doi: 10.1016/j.bbmt.2018.06.016. Epub 2018 Jun 20. PMID 29933073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multicenter study was conducted in the United States and the United Kingdom. Participants were enrolled at 5 study sites.
Pre-assignment Details: Participants with a confirmed diagnosis of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) who received an allogeneic hematopoietic stem cell transplant (HSCT) were eligible to participate and begin study drug between 42 and 84 days post HSCT. One participant was enrolled into the study but discontinued before being treated.
Groups:
- CC-486 200 mg Days 1-7 (Cohort 1): Participants received CC-486 200 mg by mouth (PO) once daily (QD) on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event (AE), disease recurrence or relapse, progressive disease (PD), development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death
- CC-486 300 mg Days 1-7 (Cohort 2): Participants received CC-486 300 mg by mouth once daily on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease, withdrawal of consent, lost to follow-up, protocol violation or death.
- CC-486 150 mg Days 1-14 (Cohort 3A): Participants received CC-486 150 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease, withdrawal of consent, lost to follow-up, protocol violation or death.
- CC-486 200 mg Days 1-14 (Cohort 3): Participants received CC-486 200 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death.
Period: Overall Study
Arm/Group | CC-486 200 mg Days 1-7 (Cohort 1) | CC-486 300 mg Days 1-7 (Cohort 2) | CC-486 150 mg Days 1-14 (Cohort 3A) | CC-486 200 mg Days 1-14 (Cohort 3)
Started (Participants who received study treatment.) | 3 | 4 | 4 | 19
Completed (Completed entire study treatment) | 1 | 0 | 2 | 10
Not Completed | 2 | 4 | 2 | 9
Not completed — Disease Recurrence or Relapse | 0 | 3 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Miscellaneous | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population includes all participants who received at least 1 dose of investigational product (IP)
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-486 200 mg Days 1-7 (Cohort 1) | CC-486 300 mg Days 1-7 (Cohort 2) | CC-486 150 mg Days 1-14 (Cohort 3A) | CC-486 200 mg Days 1-14 (Cohort 3) | Total
Number analyzed (Participants) | 3 | 4 | 4 | 19 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (5.77) | 47.8 (18.26) | 61.8 (8.73) | 60.8 (12.60) | 60.0 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 4 | 5
  Male | 2 | 4 | 4 | 15 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  White | 3 | 3 | 4 | 18 | 28
  Not Collected or Reported | 0 | 0 | 0 | 1 | 1
Diagnosis at Study Entry [Count of Participants; unit: Participants] — The number of participants with a diagnosis of AML or MDS
  Participants
    Acute Myeloid Leukemia | 2 | 4 | 4 | 16 | 26
    Myelodysplastic Syndromes | 1 | 0 | 0 | 3 | 4
MDS International Prognostic Scoring System (IPSS) Risk Classification [Count of Participants; unit: Participants] — The MDS IPSS score assesses the severity of MDS based on 3 prognostic factors each assigned a score: the percentage of bone marrow blasts, chromosome changes in the marrow cells (karyotype) and the presence of one or more low blood cell counts (cytopenias). The IPSS score is the sum of the bone marrow blast + karyotype + cytopenia score and ranges from 0 (low risk) to 3.5 (high risk). Prognosis is categorized as Low risk (score = 0), Intermediate-1 (score 0.5 to 1.0), Intermediate-2 (score 1.5 to 2.0) or High risk (score ≥ 2.5). Population: MDS Participants Have This Classification
  Participants
    number analyzed (Participants) | 1 | 0 | 0 | 3 | 4
    INT-1 | 0 | 0 | 0 | 1 | 1
    INT-2 | 1 | 0 | 0 | 1 | 2
    High | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 1 | 1 | 1 | 8 | 11
    1= Restrictive but ambulatory | 2 | 3 | 3 | 11 | 19
    2 = Ambulatory but unable to work | 0 | 0 | 0 | 0 | 0
Time from MDS or AML Diagnosis to Allogeneic HSCT [Mean (Standard Deviation); unit: months] | 8.6 (6.79) | 6.4 (4.35) | 3.5 (1.71) | 10.6 (16.72) | 8.9 (13.63)
AML World Health Organization (WHO) Classification [Number; unit: Participants:Participants] — Description:AML is classified using the WHO classification system based upon a combination of morphology, immunophenotype, genetics, and clinical features. There are several broad groups and include: 1. AML with genetic abnormalities; 2. AML with multilineage dysplasia 3. AML related to previous chemotherapy or radiation 4. Unspecified AML - do not fall into the above groups
  Participants:Participants
    AML With Recurrent Genetic Abnormalities | 0 | 2 | 0 | 7 | 9
    AML With Myelodysplasia Related Changes | 0 | 0 | 1 | 2 | 3
    Therapy related Myeloid Neoplasms | 0 | 0 | 1 | 0 | 1
    AML Not Otherwise Specified | 2 | 2 | 2 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  18-64 years | 0 | 3 | 3 | 9 | 15
  65-84 years | 3 | 1 | 1 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Dose Limiting Toxicities (DLT)
Description: A DLT included events that started within 28 days of the first dose of CC-486 in a 28-day cycle, constituted a change from baseline irrespective of outcome, as decided by the investigator to be related to CC-486 including:
  * ≥ Grade (GR) 3 nausea, diarrhea, or vomiting despite the use of medical support
  * Other significant nonhematologic toxicity of ≥ GR 3 considered not related to the disease or intercurrent illness • Absolute neutrophil count (ANC) < 0.5 x 10^9/L for > 1 week despite growth factor support
  * Platelets < 25 x 10^9/L for > 1 week despite transfusion support
  * Failure of recovery to an ANC ≥ 1.0 x 10^9/L and/or platelets ≥ 50 x 10^9/L with a hypocellular marrow by 56 days after the start of a cycle of CC-486 not due to relapse or progressive disease.
  The maximum tolerated dose is defined as the cohort delivering the highest dose in which no more than 33% of the evaluable subjects had a DLT The safety population included subjects who received ≥ 1 dose of CC-486
Time Frame: 2 months (Cycles 1 and 2)
Population: The safety population included all participants who received at least one dose of investigational product.
Measure: Number; unit: participants
Groups:
- CC-486 200 mg Days 1-7: Participants received CC-486 200 mg by mouth (PO) once daily (QD) on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event (AE), disease recurrence or relapse, progressive disease (PD), development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death
- CC-486 300 mg Days 1-7: Participants received CC-486 300 mg by mouth once daily on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease, withdrawal of consent, lost to follow-up, protocol violation or death.
- CC-486 150 mg Days 1-14: Participants received CC-486 150 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease, withdrawal of consent, lost to follow-up, protocol violation or death.
- CC-486 200 mg Days 1-14: Participants received CC-486 200 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced an adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death.
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
participants | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as any AE with an onset date on or after the first dose of IP or any event already present that worsened in severity or increased in frequency after exposure to IP up to 28 days after the last dose. In addition, an AE that occurred beyond the timeframe and was assessed by the doctor as possibly related to IP was considered to be treatment-emergent. Severity was assessed using National Cancer Institute Common Toxicity Terminology Criteria for AEs (NCI CTCAE) version 4.0, where 1= Mild; 2= Moderate; 3= Severe; 4= Life-threatening; 5= Death related to AE. Serious AEs resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in a medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes above.
Time Frame: From the first dose of investigational product (IP) up to 28 days after the last dose of IP. The median duration of exposure was 252.5 days overall; up to the final data cut off date of 14 July 2017
Population: The safety population includes all participants who received at least one dose of IP.
Measure: Number; unit: participants
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
participants
  Any TEAE | 3 | 4 | 4 | 19
  Any TEAE With A Grade 3 or 4 | 2 | 3 | 3 | 14
  Any TEAE Related to IP | 3 | 3 | 4 | 17
  TEAE With A Grade 3 or 4 Related to IP | 1 | 1 | 3 | 8
  Serious TEAE | 1 | 3 | 2 | 6
  Serious TEAE Related to IP | 1 | 0 | 1 | 2
  TEAE With Outcome of Death | 0 | 0 | 0 | 1
  TEAE Leading to Discontinuation of IP | 0 | 0 | 2 | 6
  TEAE Related to IP and Leading to Stopping IP | 0 | 0 | 1 | 3
  TEAE Leading to Dose Reduction | 0 | 0 | 0 | 1
  TEAE Leading to Dose Interruption | 1 | 0 | 1 | 6
  TEAE Leading to Dose Drug Interruption/Reduction | 0 | 0 | 0 | 1

3. Secondary Outcome: Percentage of Participants With Graft Versus Host Disease During the Entire Course of the Study
Description: Acute graft versus host disease generally occurs after allogeneic hematopoietic stem cell transplantation. It is a reaction of donor immune cells against host tissues. The 3 main tissues that acute GVHD affects are the skin, liver, and gastrointestinal tract. Chronic GVHD is scored per the National Institute of Health consensus conference grading system. Clinical manifestations of chronic GVHD include skin involvement resembling lichen planus or the cutaneous manifestations of scleroderma; dry oral mucosa with ulcerations and sclerosis of the gastrointestinal tract; and a rising serum bilirubin concentration.
Time Frame: From the first dose of CC-486 up to study discontinuation or death. Up to final data cut off date of 14 July 2017; up to 186 weeks and 4 days
Population: Safety population includes all participants who received at least 1 dose of IP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CC-486 200 mg Days 1-7: Participants received CC-486 200 mg by mouth (PO) once daily (QD) on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced, adverse event (AE), disease recurrence or relapse, progressive disease (PD), development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death
- CC-486 200 mg Days 1-14: Participants received CC-486 200 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced, adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death.
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
percentage of participants | 66.7 [9.43 to 99.16] | 0.0 [0.00 to 60.24] | 75.0 [19.41 to 99.37] | 63.2 [38.36 to 83.71]

4. Secondary Outcome: Kaplan Meier Estimate of Time to Discontinuation From Treatment
Description: The time to discontinuation from treatment was assessed as an estimate of treatment tolerability and was defined as the interval from the date of the first IP dose to the date of discontinuation from IP as indicated on the discontinuation from treatment Case Report Form page. Time to discontinuation from study treatment was analyzed using the Kaplan-Meier method where participants who did not discontinue were censored at the date of last visit.
Time Frame: From the first dose of IP dose to the date of discontinuation from IP; the overall median time to discontinuation of IP was 283.5 days
Population: The safety population includes all participants who received at least one dose of investigational product. Participants who were on treatment at the time of study closure were censored at the date of last available visit
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
Days | 189.0 [184.0 to NA] — NA indicates time was not reached due to participants remaining in study until study closure. | 177.0 [104.5 to 189.0] | NA [228.5 to NA] — NA indicates time was not reached due to participants remaining in study until study closure | 389.0 [58.0 to NA] — NA indicates time was not reached due to participants remaining in study until study closure

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration Of CC-486 (AUC-t)
Description: Area under the plasma concentration-time curve from Time 0 to the time of the last quantifiable concentration, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: On Day 1, pharmacokinetic (PK) samples were collected at predose and over a 6-hour period following drug administration on the following schedule: 0.5, 1, 1.5, 2, 2.5, 3, 4, and 6 hours post-dose; Cycle 1 or 2 until 6 hours after CC-486 administration.
Population: The PK population were those with evaluable CC-486 plasma PK profiles; PK data from those who received CC-486 200 mg QD were combined because following a single CC-486 dose, the half-life elimination is <1 h; CC 486 does not accumulate following multiple administrations. CC-486 200 mg Days 1-7 and CC-486 200 mg Days 1-14 arms can be combined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- CC-486 200 mg Days 1-7 and Days 1-14: Pharmacokinetic data from participants who received CC-486 200 mg by mouth daily were combined because the wash-out period between the PK sample collection and previous CC-486 dose was greater than 7-fold the half-life elimination of the drug, and CC 486 does not accumulate following multiple administrations.
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 20 | 5 | 2
ng*h/mL
  Without Concomitant Meds: number analyzed (Participants) | 4 | 2 | 0
  Without Concomitant Meds | 204.6 (63.0) | 253.3 (26.6) |
  With Concomitant Meds | 176.8 (69.0) | 226.7 (54.5) | 187.2 (34.19)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Extrapolated to Infinity (AUC-inf; AUC0-∞) Of CC-486
Description: Area under the plasma concentration-time curve from time 0 extrapolated to infinity, calculated as [AUCt + Ct/ λz]. Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz. If AUC %Extrap was ≥25%, AUC inf was not reported.
Time Frame: On Day 1, PK samples were collected at predose and over the 6-hour period following CC-486 administration on the following schedule: 0.5, 1, 1.5, 2, 2.5, 3, 4, and 6 hours post-dose at Cycle 1 or 2 until 6 hours after CC-486 administration.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 18 | 5 | 2
ng*h/mL
  Without Concomitant Meds: number analyzed (Participants) | 4 | 1 | 0
  Without Concomitant Meds | 206.0 (62.8) | 218.4 (NA) — Could not be calculated as sample size = 1. |
  With Concomitant Meds | 187.5 (70.1) | 232.5 (51.7) | 188.6 (33.5)

7. Secondary Outcome: Maximum Observed Concentration (Cmax) Of CC-486
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 20 | 5 | 2
ng/mL
  Without Concomitant Meds: number analyzed (Participants) | 4 | 2 | 0
  Without Concomitant Meds | 151.9 (43.59) | 149.8 (7.6) |
  With Concomitant Meds | 114.3 (73.4) | 137.85 (65.7) | 91.49 (25.1)

8. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of CC-486
Description: Time to Cmax, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- CC-486 200 mg Days 1-7 and Days 1-14-day: Pharmacokinetic data from participants who received CC-486 200 mg by mouth daily were combined because the wash-out period between the PK sample collection and previous CC-486 dose was greater than 7-fold the half-life elimination of the drug, and CC 486 does not accumulate following multiple administrations.
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14-day | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 20 | 5 | 2
hours
  Without Concomitant Meds: number analyzed (Participants) | 4 | 2 | 0
  Without Concomitant Meds | 0.77 [0.50 to 1.5] | 2.3 [1.5 to 3.1] |
  With Concomitant Meds | 1.5 [0.47 to 3.0] | 2.0 [1.5 to 2.5] | 2.0 [2.0 to 2.0]

9. Secondary Outcome: Terminal Half-Life (T1/2) of CC-486
Description: Terminal phase half-life in plasma, calculated as [(ln 2)/λz]. t1/2 will only be calculated when a reliable estimate for λz can be obtained.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 18 | 5 | 2
hours
  Without Concomitant Meds: number analyzed (Participants) | 4 | 1 | 0
  Without Concomitant Meds | 0.528 (6.8) | 0.575 (NA) — Could not be calculated since sample size = 1 |
  With Concomitant Meds | 0.553 (24.5) | 0.565 (44.3) | 0.446 (20.6)

10. Secondary Outcome: Apparent Total Clearance (CL/F) of CC-486
Description: Apparent total clearance, calculated as [Dose/AUCinf].
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- CC-486 200 mg Days 1-7 and Day 1-14: Pharmacokinetic data from participants who received CC-486 200 mg by mouth daily were combined because the wash-out period between the PK sample collection and previous CC-486 dose was greater than 7-fold the half-life elimination of the drug, and CC 486 does not accumulate following multiple administrations.
Arm/Group | CC-486 200 mg Days 1-7 and Day 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 18 | 5 | 2
L/h
  Without Concomitant Meds: number analyzed (Participants) | 4 | 1 | 0
  Without Concomitant Meds | 971.1 (62.8) | 1374 (NA) — Could not be calculated since sample size = 1 |
  With Concomitant Meds | 1067 (70.1) | 1290 (51.7) | 795.4 (33.5)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of CC-486
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | CC-486 200 mg Days 1-7 and Days 1-14 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14
Number analyzed (Participants) | 18 | 5 | 2
Liters
  Without Concomitant Meds: number analyzed (Participants) | 4 | 1 | 0
  Without Concomitant Meds | 739.9 (58.7) | 1139 (NA) — Could not be calculated since sample size = 1 |
  With Concomitant Meds | 851.3 (77.6) | 1052 (100.0) | 511.8 (12.3)

12. Secondary Outcome: Percentage of Participants With Disease Relapse or Progression
Description: Disease relapse was defined as the reappearance of > 5% blasts in the bone marrow that persists for at least 4 weeks. Disease progression was defined as the reappearance of > 10% of blasts in the bone marrow that persisted for at least 4 weeks.
Time Frame: Date of first dose of IP to disease relapse or progression; up to data cut-off date of 14 July 2017; median number of days assessed was 963.0 days for Cohort 1, 743.5 days for Cohort 2, 675.5 days for Cohort 3A and 559.0 days for Cohort 3.
Population: Preliminary efficacy population included all participants who received at ≥ 1 dose of IP and had at ≥ 1 post-baseline efficacy assessment performed.
Measure: Number; unit: Percentage of Participants
Groups:
- CC-486 200 mg Days 1-7 (Cohort 1): Participants received CC-486 200 mg by mouth (PO) once daily (QD) on Days 1 to 7 of each 28-day cycle for a maximum duration of 12 months or until they experienced, adverse event (AE), disease recurrence or relapse, progressive disease (PD), development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death
- CC-486 200 mg Days 1-14 (Cohort 3): Participants received CC-486 200 mg by mouth once daily on Days 1 to 14 of each 28-day cycle for a maximum duration of 12 months or until they experienced, adverse event, disease recurrence or relapse, progressive disease, development of Grade III/IV acute graft versus host disease (GVHD), withdrawal of consent, lost to follow-up, protocol violation or death.
Arm/Group | CC-486 200 mg Days 1-7 (Cohort 1) | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14 (Cohort 3)
Number analyzed (Participants) | 3 | 4 | 4 | 19
Percentage of Participants | 33.3 | 75.0 | 0 | 15.8

13. Secondary Outcome: Time to Disease Recurrence/Progression
Description: Time to disease relapse/progression was defined as the interval from the date of allogeneic HSCT to the date of treatment discontinuation or study discontinuation where reason for discontinuation is disease relapse or disease progression, or the date of disease progression recorded on the survival electronic Case Report Form page, whichever occurred first. Time to disease relapse/progression was analyzed using competing risk methods where death without documented relapse/progression was treated as a competing risk for relapse/progression. relapse/progression.
Time Frame: Date of allogenic HSCT to disease progression or relaopse; up to data cut-off date of 14 July 2017; median number of days assessed was 963.0 days for Cohort 1, 743.5 days for Cohort 2, 675.5 days for Cohort 3A and 559.0 days for Cohort 3.
Population: Preliminary efficacy population included all participants who received at ≥ 1 dose of IP and had at ≥ 1 post-baseline efficacy assessment performed. Participants who were lost to follow-up without documented relapse/progression, or were alive at last follow-up without documented relapse/progression were censored at the date of the last assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
days | 691.7 (436.10) | 452.5 (493.50) | 660.8 (218.12) | 521.7 (310.53)

14. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from the date of allogeneic hematopoietic stem cell transplantation to death from any cause.
Time Frame: Date of the allogeneic HSCT to death from any cause. Median number of days participants were assessed from first dose to last contact was 963.0 days for Cohort 1, 743.5 days for Cohort 2, 675.5 days for Cohort 3A and 559.0 days for Cohort 3.
Population: Preliminary efficacy population includes all participants who received at least 1 dose of IP and had at least 1 post-baseline efficacy assessment performed. All participants were followed until drop-out, death, or study closure. Participants who dropped out or were alive at study closure were censored at the time of last contact, as appropriate.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
Days | NA [741.0 to NA] — NA as OS was not reached due to long survival of subjects relative to study duration. | NA [303.5 to NA] — NA as OS was not reached due to long survival of subjects relative to study duration. | NA [NA to NA] — NA as OS was not reached due to long survival of subjects relative to study duration. | NA [467.0 to NA] — NA as OS was not reached due to long survival of subjects relative to study duration.

15. Secondary Outcome: Kaplan Meier Estimate of Relapse-Free Survival (RFS)
Description: Relapse-free survival was defined as the interval from the date of allogeneic HSCT to the date of first documented > 5% blasts in the bone marrow or death from any cause, whichever occurs first. Participants who were still alive and continued to have less than or equal to 5% blasts in the bone marrow or who were lost to follow-up were censored at the date of their last response assessment.
Time Frame: Date of allogenic HSCT to date of progression or death from any cause; Median number of days participants were assessed from first dose to last contact was 963 days for Cohort 1, 674.8 days for Cohort 2, 577.5 days for Cohort 3A and 553 days for Cohort 3
Population: Preliminary efficacy population includes all participants who received at least 1 dose of IP and had at least 1 post-baseline efficacy assessment performed. Participants who were still alive and continued to have ≤5% blasts in the bone marrow or who were lost to follow-up were censored at the date of their last response assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | CC-486 200 mg Days 1-7 | CC-486 300 mg Days 1-7 | CC-486 150 mg Days 1-14 | CC-486 200 mg Days 1-14
Number analyzed (Participants) | 3 | 4 | 4 | 19
Days | 921.0 [741.0 to 1101.0] | 255.0 [183.0 to NA] — NA as RFS was not reached due to long survival of subjects relative to study duration. | NA [NA to NA] — NA as RFS was not reached due to long survival of subjects relative to study duration. | NA [281.0 to NA] — NA as RFS was not reached due to long survival of subjects relative to study duration.

ADVERSE EVENTS:
Time Frame: From the first dose of IP up to 28 days after the last dose of IP. The median duration of exposure was 252.5 days overall.
Arm/Group | CC-486 200 mg Days 1-7 (Cohort 1) | CC-486 300 mg Days 1-7 (Cohort 2) | CC-486 150 mg Days 1-14 (Cohort 3A) | CC-486 200 mg Days 1-14 (Cohort 3)
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/4 | 2/4 | 11/19
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 2/4 | 6/19
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 200 mg Days 1-7 (Cohort 1) (N=3) | CC-486 300 mg Days 1-7 (Cohort 2) (N=4) | CC-486 150 mg Days 1-14 (Cohort 3A) (N=4) | CC-486 200 mg Days 1-14 (Cohort 3) (N=19)
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 0 | 0 | 3
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-486 200 mg Days 1-7 (Cohort 1) (N=3) | CC-486 300 mg Days 1-7 (Cohort 2) (N=4) | CC-486 150 mg Days 1-14 (Cohort 3A) (N=4) | CC-486 200 mg Days 1-14 (Cohort 3) (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 6
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 12
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 8
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 2 | 7
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 2
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 0 | 1 | 2
Graft versus host disease in liver (Immune system disorders) | 0 | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Corneal infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 4
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 3
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission up to 90 additional days. Investigator must delete confidential data before submission or defer publication to permit patent applications.